CLINICAL TRIAL: NCT04883593
Title: A Multi-center, Double-blind, Randomized, Placebo Controlled, Parallel-Group Study, Comparing TA103 and Placebo Control in the Treatment of Tinea Pedis.
Brief Title: A Study Comparing the Efficacy of TA103 and the Placebo Control in the Treatment of Interdigital Tinea Pedis.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TA103-2004
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TA103 (Experimental): The assigned Investigational Product will be applied to the skin between, under, all over the toes, sole and sides of the entire foot. Both feet are to be treated in the same way, even if the skin looks healthy and lesions are present on one foot only.
  Interventions: Drug: TA103
- Placebo Control (Placebo Comparator): The assigned Investigational Product will be applied to the skin between, under, all over the toes, sole and sides of the entire foot. Both feet are to be treated in the same way, even if the skin looks healthy and lesions are present on one foot only.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: TA103 — The assigned Investigational Product will be applied to the skin between, under, all over the toes, sole and sides of the entire foot. Both feet are to be treated in the same way, even if the skin looks healthy and lesions are present on one foot only.
  Other Names: Test Product
  Arms: TA103
Drug: Placebo Control — The assigned Investigational Product will be applied to the skin between, under, all over the toes, sole and sides of the entire foot. Both feet are to be treated in the same way, even if the skin looks healthy and lesions are present on one foot only.
  Other Names: Vehicle
  Arms: Placebo Control

SUMMARY:
To evaluate and compare the safety and efficacy of TA103 in the treatment of tinea pedis.

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, placebo controlled, parallel-group study, comparing TA103 and the placebo control in the treatment of tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 18 years
* Subjects must have provided IRB approved written informed consent
* Subjects must have clinical diagnosis of interdigital tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot (the non-interdigital lesions should not be hyperkeratotic, i.e., characteristic of tinea pedis moccasin).

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Subjects with a history of hypersensitivity or allergy to any of the study medication ingredients and its excipients.
* Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with complete cure at Week 6 (+/- 4 days) following treatment (study day 38-46) | Baseline to Week 6 Visit
  To evaluate safety and efficacy of TA103

CONTACTS AND LOCATIONS:
Overall Officials: Zaidoon A. Al-Zubaidy, Study Director — Catawba Research
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States